CLINICAL TRIAL: NCT07404579
Title: A Phase II, Multicenter, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Efficacy and Safety of Bolus-Administered HRS-9190 Versus Rocuronium for Maintaining Neuromuscular Blockade During General Anesthesia in Adults Undergoing Elective Surgery.
Brief Title: Safety and Efficacy of HRS-9190 Compared to Rocuronium for Bolus Maintenance in Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9190-202
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment group A: HRS-9190 under Inhalational Anesthesia (Experimental)
  Interventions: Drug: HRS-9190
- Treatment group B: HRS-9190 under Inhalational Anesthesia (Experimental)
  Interventions: Drug: HRS-9190
- Treatment group C: HRS-9190 under Intravenous Anesthesia (Experimental)
  Interventions: Drug: HRS-9190
- Treatment group D: HRS-9190 under Intravenous Anesthesia (Experimental)
  Interventions: Drug: HRS-9190
- Treatment group E: Rocuronium under Inhalational Anesthesia (Active Comparator)
  Interventions: Drug: Rocuronium
- Treatment group F: Rocuronium under Intravenous Anesthesia. (Active Comparator)
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: HRS-9190 — HRS-9190; high dose(under Inhalational Anesthesia)
  Arms: Treatment group A: HRS-9190 under Inhalational Anesthesia
Drug: HRS-9190 — HRS-9190; low dose(under Inhalational Anesthesia)
  Arms: Treatment group B: HRS-9190 under Inhalational Anesthesia
Drug: HRS-9190 — HRS-9190; high dose(under Intravenous Anesthesia)
  Arms: Treatment group C: HRS-9190 under Intravenous Anesthesia
Drug: HRS-9190 — HRS-9190; low dose(under Intravenous Anesthesia)
  Arms: Treatment group D: HRS-9190 under Intravenous Anesthesia
Drug: Rocuronium — Rocuronium(under Inhalational Anesthesia).
  Arms: Treatment group E: Rocuronium under Inhalational Anesthesia
Drug: Rocuronium — Rocuronium(under Intravenous Anesthesia)
  Arms: Treatment group F: Rocuronium under Intravenous Anesthesia.

SUMMARY:
The study will enroll adult patients scheduled for elective surgery requiring general anesthesia. Participants will be randomly assigned to receive either HRS-9190 for Injection or Rocuronium. The primary objective is to measure the duration from the last dose of the study drug until the recovery of neuromuscular function to a specific level (TOFr ≥ 90%). Secondary objectives include evaluating the onset time and duration of action following each dose, the total time adequate muscle relaxation is maintained during surgery, and the detailed pattern of neuromuscular recovery. Safety assessments will include monitoring of adverse events, vital signs, laboratory parameters, and other safety indicators throughout the study period. The hypothesis of this study is that HRS-9190 for Injection could provide effective neuromuscular relaxation, with a satisfied safety profile in the target patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia surgery
3. Meet specified age and body mass index (BMI) criteria
4. Conform to the ASA Physical Status Classification
5. Use of highly effective contraception for a specified period if applicable

Exclusion Criteria:

1. Scheduled for specific high-risk surgical procedures
2. History of significant neuromuscular, cardiovascular, respiratory, or neurological disorders
3. History of conditions affecting drug metabolism or anesthesia risk
4. Abnormal laboratory values indicating significant clinical abnormalities
5. Positive serology for specified infectious diseases
6. Known hypersensitivity to related medications
7. Recent use of medications interfering with neuromuscular function
8. History of mental illness, cognitive impairment, or epilepsy
9. Participation in another clinical trial within a specified period
10. Any other condition deemed unsuitable by the investigator
11. Pregnant or nursing women
12. Unwilling to use birth control during the specified period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time from Last Dose to Recovery of TOFr to 0.9 | From the administration of the last dose of the study drug until TOFr ≥ 0.9 is achieved, assessed intraoperatively and in the recovery period, up to 2 hours.
  The duration (in minutes) from the administration of the last dose of the neuromuscular blocking agent to the recovery of the Train-of-Four ratio (TOFr) to 90% or greater

SECONDARY OUTCOMES:
Duration of Action after Bolus Dose(s) | For each bolus dose: from administratin until specified recovery points, assessed intraoperatively, up to 2 hours.
  The time (in minutes) from each bolus administration (including the initial dose for induction) to: 1) the start of T1 recovery; 2) recovery of T1 to 10% of baseline; 3) recovery of T1 to 25% of baseline.
Time from Last Dose to Specific TOFr Recovery Milestones | From the administration of the last dose of the study drug until specified TOFr values are achieved, assessed intraoperatively and in recovery, up to 2 hours.
  The time (in minutes) from the last dose to the recovery of TOFr to 0.4 and to 0.7.
Percentage of Time with Target Neuromuscular Block | From the first administration of the study drug until the end of the last maintenance dose requirement, assessed intraoperatively, up to 6 hours.
  The proportion (%) of the total drug administration period during which adequate surgical relaxation (T1 ≤ 25% of baseline) is maintained.
Time to Successful Airway Device Placement | From administration of the initial intubating dose to completion of tracheal intubation or laryngeal mask insertion, assessed at induction, approximately 2-5 minutes.
  The time (in minutes) from the administration of the study drug for induction to the completion of tracheal intubation or laryngeal mask placement.
Onset Time after Bolus Dose(s) | For each bolus dose: from administration to maximum T1 depression, assessed intraoperatively, up to 6 hours.
  The time (in minutes) from each bolus administration (including for induction) to the time of maximum T1 depression (peak effect).
Time from Last Dose to Airway Device Removal | From the administration of the last dose of the study drug to tracheal extubation or laryngeal mask removal, assessed at the end of surgery until device removal, up to 2 hours.
  The time (in minutes) from the last dose of the study drug to the removal of the tracheal tube or laryngeal mask.
Recovery Index | After the last dose: from T1=25% to T1=75%, and from T1=5% to T1=95%, assessed intraoperatively and in recovery, up to 2 hours.
  The recovery time (in minutes) for T1 to recover from 25% to 75% of baseline, and from 5% to 95% of baseline, following the last dose.
Anesthesiologist's Overall Satisfaction Score | Assessed at the end of the surgical procedure, within 1 hour.
  The overall satisfaction score regarding the quality and ease of neuromuscular management, rated by the attending anesthesiologist using a predefined scale.
Surgeon's Overall Satisfaction Score | Assessed at the end of the surgical procedure, within 1 hour.
  The overall satisfaction score regarding surgical conditions related to muscle relaxation, rated by the operating surgeon using a predefined scale.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided